CLINICAL TRIAL: NCT03510546
Title: Effect of Pyridostigmine (Mestinon) on Muscle Strength in Myasthenia Gravis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Jan Lykke Scheel Thomsen, MD, PhD Fellow, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Mestinon2018
Record Dates: First submitted 2018-04-06; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Pyridostigmine Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): De-novo: Each capsule contains 60 mg. pyridostigmine. 1 capsule is administered twice within 4 hours.
  Chronic: Each capsule contains 60 mg. pyridostigmine. Number of administered capsules per dosage depend on the patient's usual dosage. Study drug is administered twice within 4 hours.
  Patients are examined/rated before 1st dose, 1 hour after 1st dose, 1 hour after 2nd dose (Visit 1). After cross-over (Visit 2), patients will be rated open-label at 1 month (Visit 3) and 3 months (Visit 4).
  Interventions: Drug: Pyridostigmine
- Placebo (Placebo Comparator): Same as "Active", however capsules contain placebo.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Pyridostigmine — Study dose as per protocol.
  Arms: Active
Drug: Placebo oral capsule — Study dose as per protocol.
  Arms: Placebo

SUMMARY:
A randomized, placebo-controlled, double-blinded cross-over study evaluating and quantifying the effect of pyridostigmine on muscle strength and symptoms in Myasthenia Gravis (MG)

DETAILED DESCRIPTION:
The study aims to evaluate and quantify the effect of pyridostigmine on symptoms and muscle strength in newly-diagnosed patients and patients on stable medication.

Pyridostigmine treatment is initiated in the vast majority of MG patients. No studies have quantified the effect in a randomized trial, and no studies have examined the potential difference in effect in newly diagnosed patients as compared to patients on stable, antimyasthenic medications.

The study will investigate the effect in two groups

1. Newly diagnosed, treatment-naive patients.
2. MG patients on stable antimyasthenic medication.

ELIGIBILITY:
Inclusion Criteria:

* MG verified by a) anti-body, or b) single-fiber EMG and/or decrement on ENG.

Exclusion Criteria:

* Anti-MuSK
* Known cardio-pulmonary disease
* Known neuropathy
* Known myopathy
* Known malignant disease
* Pregnancy or breastfeeding
* Mechanic ileus, urinary tract obstruction, peritonitis

De-novo MG Eligibility Criteria

* MG diagnosis < 2 months, no prior antimyasthenic medications

Chronic MG Eligibility Criteria

* MG diagnosis > 1 year, and stable pyridostigmine dosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-04-09 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in QMG | At baseline, 1 hour after 1st dose (administered immediately after baseline assessment), 1 hour after 2nd dose (administered 2 hours after 1st dose). Assessed on Day 1 and Day 2 (cross-over), at Follow-up 1 (1 month) and Follow-up 2 (3 months).
  Quantitative Myasthenia Gravis (QMG) scale rate disease severity of myasthenia gravis on 13 items with a total score ranging from 0-39 (higher values representing more severe disease). Total score (0-39), ocular subitems (0-6), bulbar subitems (0-9), extremity/axial subitems (0-21) and respiratory subitem (0-3) will be reported.

SECONDARY OUTCOMES:
Change in muscle strength as assessed by dynamometry (Biodex System 3). | At baseline, 1 hour after 1st dose (administered immediately after baseline assessment), 1 hour after 2nd dose (administered 2 hours after 1st dose). Assessed on Day 1 and Day 2 (cross-over), at Follow-up 1 (1 month) and Follow-up 2 (3 months).
  Peak muscle torque expressed in newton meters based on 3 repeated maximal isometric contractions. Performed on shoulder abduction and knee extension.
Change in muscle fatigue as assessed by dynamometry (Biodex System 3). | At baseline, 1 hour after 1st dose (administered immediately after baseline assessment), 1 hour after 2nd dose (administered 2 hours after 1st dose). Assessed on Day 1 and Day 2 (cross-over), at Follow-up 1 (1 month) and Follow-up 2 (3 months).
  Decrement in peak muscle torque expressed in newton meters per contraction during up to 50 repetitive maximal isokinetic contractions. Performed on shoulder abduction and knee extension.
Change in MG Composite Score | At baseline, 1 hour after 1st dose (administered immediately after baseline assessment), 1 hour after 2nd dose (administered 2 hours after 1st dose). Assessed on Day 1 and Day 2 (cross-over), at Follow-up 1 (1 month) and Follow-up 2 (3 months).
  The Myasthenia Gravis Composite (MG composite) scale rate disease severity of myasthenia gravis on 10 items with a score ranging from 0-50 (higher values representing more severe disease).

CONTACTS AND LOCATIONS:
Overall Officials: Jan LS Thomsen, MD, Principal Investigator — University of Aarhus
Locations (1):
- Department of Neurology Aarhus University Hospital, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnett C, Katzberg H, Nabavi M, Bril V. The quantitative myasthenia gravis score: comparison with clinical, electrophysiological, and laboratory markers. J Clin Neuromuscul Dis. 2012 Jun;13(4):201-5. doi: 10.1097/CND.0b013e31824619d5. PMID 22622164
- [Background] Burns TM, Conaway M, Sanders DB; MG Composite and MG-QOL15 Study Group. The MG Composite: A valid and reliable outcome measure for myasthenia gravis. Neurology. 2010 May 4;74(18):1434-40. doi: 10.1212/WNL.0b013e3181dc1b1e. PMID 20439845